CLINICAL TRIAL: NCT05118854
Title: A Phase II Study of Neoadjuvant Sotorasib in Combination With Cisplatin or Carboplatin and Pemetrexed for Surgically Resectable Stage IIA-IIIB Non-Squamous Non-Small Cell Lung Cancer With a KRAS p.G12C Mutation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0649; NCI-2021-10907 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2021-09-28; First posted 2021-11-12 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — sotorasib; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sotorasib in Combination with Cisplatin/Carboplatin and Pemetrexed (Experimental): 4 cycles of at least one dose of sotorasib plus cisplatin (or carboplatin) and pemetrexed can be administered safely
  Interventions: Drug: AMG 510; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: AMG 510 — Given by IV
Drug: Cisplatin — Given by IV
  Other Names: Platinol®-AQ; Platinol®; CDDP
Drug: Carboplatin — Given by IV
Drug: Pemetrexed — Given by IV
  Other Names: LY231514; Alimta®; MTA; Multitargeted Antifolate; NSC-698037

SUMMARY:
This is a phase II, single-arm, open-label study evaluating the efficacy, safety and tolerability of neoadjuvant sotorasib in combination with cisplatin (or carboplatin) and pemetrexed chemotherapy for patients with surgically resectable stage IIA - IIIB (T3-T4/N2) (based on AJCC 8th edition), non-squamous NSCLC with a KRAS p.G12C mutation. The primary objective of the study is to determine whether neoadjuvant therapy with 4 cycles of at least one dose of sotorasib plus cisplatin (or carboplatin) and pemetrexed can be administered safely and result in improved MPR rate in patients with KRAS p.G12C-mutant non-squamous NSCLC compared with the historical control MPR rate for platinum-based chemotherapy alone.

DETAILED DESCRIPTION:
Objectives

Primary:

* To evaluate the efficacy of induction with sotorasib (AMG 510) in combination with cisplatin (or carboplatin) and pemetrexed in patients with surgically resectable KRAS p.G12C-mutant non-squamous NSCLC as assessed by major pathologic response rate in resected tumor specimens.
* To determine the safety, tolerability and RP2D of sotorasib in combination with cisplatin (or carboplatin) and pemetrexed as induction therapy in patients with surgically resectable KRAS p.G12C-mutant nonsquamous NSCLC

Secondary:

* To evaluate the efficacy of induction sotorasib in combination with cisplatin (or carboplatin) and pemetrexed in patients with surgically resectable KRAS p.G12C mutant non-squamous NSCLC as assessed by : Objective response rate (ORR), Eventfree survival, Recurrence-free survival, Overall Survival (OS), Complete Resection (R0) and Pathologic complete response rate (pCR)
* To determine the safety and tolerability of sotorasib in combination with cisplatin (or carboplatin) and pemetrexed as induction therapy in patients with surgically resectable KRAS p.G12C-mutant nonsquamous NSCLC.

Exploratory:

* To evaluate biomarkers of response to induction sotorasib in combination with cisplatin (or carboplatin) and pemetrexed in surgically resectable KRAS p.G12C-mutant non-squamous NSCLC.
* To assess modulation of tissue and/or blood markers in response to induction with sotorasib in combination with cisplatin (or carboplatin) and pemetrexed in surgically resectable KRAS p.G12C-mutant nonsquamous NSCLC.
* To evaluate mechanisms of adaptation and/or resistance to sotorasib in combination with cisplatin (or carboplatin) and pemetrexed in surgically resectable KRAS p.G12C-mutant non-squamous NSCLC.
* To evaluate immune modulation in tissue and the periphery in response to induction sotorasib in combination with cisplatin (or carboplatin) and pemetrexed in surgically resectable KRAS p.G12C-mutant nonsquamous NSCLC.

ELIGIBILITY:
Inclusion Criteria

1. [*] Subject or subject's legally acceptable representative has provided signed and dated written informed consent prior to initiation of any study specific activities/procedures in accordance with ICH-GCP guidelines and the local legislation.
2. [*]Age > 18 years old.
3. [*]Histologically or cytologically confirmed previously untreated non-squamous non-small cell lung cancer. If a diagnostic biopsy is available, a pre-treatment biopsy is not required. Patients with a suspected lung cancer are eligible, but pathology must be confirmed prior to initiating treatment on study. Pure squamous cell carcinomas are not eligible but mixed histologies (for example adenosquamous carcinoma) are eligible. Sarcomatoid carcinomas are not eligible.

   Neuroendocrine carcinomas are not eligible. Carcinomas with neuroendocrine differentiation are eligible. Patients with mixed small-cell lung cancer and NSCLC are not eligible.
4. Identification of a KRAS p.G12C mutation in tumor tissue or plasma by an approved diagnostic device for detection of KRAS p.G12C in NSCLC or through any nucleic acid-based diagnostic testing method [including droplet-digital PCR, real-time PCR based methods such as the Idylla KRAS Mutation Assay (Biocartis), tissue and circulating tumor DNA -based next generation sequencing, Sanger-sequencing etc] performed in a Clinical Laboratory Improvement Amendments (CLIA)-certified or equivalently accredited laboratory. Patients meeting [*] highlighted criteria will be offered study-provided droplet digital PCR or alternative PCR-based method such as the Idylla KRAS Mutation Assay (Biocartis) for detection of KRAS p.G12C using tumor tissue (1st choice if adequate tissue is available) or plasma (if tumor tissue is not available or cannot be accessed within 5 working days). Turnaround time for reporting of the presence or absence of a KRAS p.G12C mutation will be ≤ 5 working daysfor plasma-based testing and ≤7 working days from the date of confirmation of tissue availability for tissue-based testing. If analysis of tumor tissue fails due to technical reasons, the same patient can undergo analysis of circulating tumor DNA using droplet-digital PCR or alternative PCR-based method such as the Idylla KRAS Mutation Assay (Biocartis). If plasma-based analysis failes to detect a KRAS p.G12C mutation and tumor tissue becomes available, the same patient can undergo analysis of tumor tissue using droplet digital PCR or alternative PCR-based method such as the Idylla KRAS Mutation Assay (Biocartis).
5. Patients with disease stage IIA to select stage IIIB (T3-4N2) (according to version 8 of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology [IASLC Staging Manual in Thoracic Oncology 2016]). Patients with multistation N2 disease are eligible provided that complete surgical resection is considered feasible by multidisciplinary evaluation which must include a thoracic surgeon that performs lung cancer surgery as a prominent part of his/her practice Invasive mediastinal staging with endosonography (EBUS or EUS) with fine-needle aspiration (FNA) and/or mediastinoscopy should be completed within 42 days from the start of treatment in the following cases:

   * In case of mediastinal lymph nodes that are enlarged by CT criteria and/or PET-positive mediastinal lymph nodes.
   * In case of tumors > 3 cm in maximum diameter
   * In case of centrally located tumors
   * For tumors with N1 nodes (cN1) Invasive mediastinal staging should include evaluation of contralateral stations 2 and/or 4 to exclude N3 disease as well as of subcarinal (station 7) lymph nodes. When there are no enlarged mediastinal lymph nodes by CT criteria and there is no uptake on PET/CT (cN0) direct surgical resection with lymph node dissection is indicated for tumors ≤ 3cm that are located in the outer third of the lung.
6. [*] Absence of unequivocal evidence of stage IV disease based on contrast-enhanced CT chest, abdomen, pelvis or PET/CT and brain MRI with IV contrast (or contrast-enhanced CT of the head) performed within 60 days is sufficient for study registration but must be confirmed with whole-body PET/CT as well as contrast-enhanced CT chest and abdomen (or contrast-enhanced CT chest including the whole liver and both adrenal glands) and brain MRI with IV contrast (or contrast-enhanced CT of the head) within 28 days prior to the start of treatment. Patients with lesions that are considered equivocal for metastatic disease in the opinion of the local principal investigator are elibile to register and undergo molecular testing if they meet all other [*] marked criteria but must meet the full trial eligibility criteria prior to study enrollment. In patients with severe allergy to iodinated contrast absence of stage IV disease on PET/CT and brain MRI with IV contrast performed within 28 days prior to enrollment suffices to satisfy this eligibility criterion.
7. [*]Measurable disease based on RECIST 1.1 as determined by the local site investigator/radiology assessment.
8. [*]The patient must be a suitable candidate for surgery, in the opinion of the treating physician.
9. [*]ECOG performance status score 0-1and life expectancy > 3 months (in the opinion of the investigator).
10. [*]Patients must be able to take oral medications and willing to record daily adherence to investigational product.
11. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≤ 470 msec in females and QTcF ≤ 450 msec in males (based on average of screening triplicates performed within 5 minutes).
12. Subjects must have available (or accessible) and be willing to provide archival tumor tissue samples (formalin-fixed paraffin-embedded [FFPE] sample [FFPE of excisional biopsy, core needle biopsy or fine needle aspirates] collected within 5 years) or be willing to undergo pretreatment tumor biopsy (excisional, core needle, or fine needle aspirates) prior to enrollment.

    Subjects who do not have archived tissue available can be allowed to enroll without undergoing tumor biopsy upon agreement with the overall study PI if a tumor biopsy is not feasible.
13. Patients must have adequate hematologic laboratory assessments, defined as the following within 10 days prior to start of study therapy:

    1. Absolute neutrophil count (ANC) ≥ 1500 cells/µl (without granulocyte colony-stimulating factor support within 10 days of laboratory test used to determine eligibility).
    2. Hemoglobin ≥ 9.0 g/dL (without transfusion within 2 weeks of laboratory test used to determine eligibility).
    3. Platelet count ≥ 100,000/µl (without transfusion within 2 weeks of laboratory test used to determine eligibility).
14. Prothrombin time (PT)≤1.5 x ULN or International normalized ratio (INR) ≤1.5 x ULN (or within the target range if on prophylactic anticoagulation therapy) and (activated) partial thromboplastin time (PTT or aPTT)≤1.5 x ULN unless the patient is receiving therapeutic anticoagulation in which case they should be within therapeutic target limits.
15. Patients must have adequate liver function, defined as the following:

    1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN), except if alkaline phosphatase > 2.5 times the ULN in which case AST and/or ALT must be ≤ 1.5 times the ULN.
    2. Serum bilirubin ≤ 1.0 x ULN, except in subjects with Gilbert Syndrome, who can have total bilirubin < 2.0 mg/dL.
16. Subjects must have calculated creatinine clearance ≥ 60 mL/min (based on the Cockroft-Gault formula1 ), using actual body weight. Twenty-four hour urine collection for calculation of creatinine clearance is not required but is allowed

Exclusion Criteria:

1. [*]Current or prior systemic anticancer therapy (chemotherapy, immunotherapy, biological therapy, hormonal therapyor other investigational anti-cancer drug) or radiation therapy for treatment of the current lung cancer. Concurrent use of hormonal therapy for non-cancer-related conditions (such as hormone replacement therapy) is allowed.
2. [*]Pure squamous or predominantly squamous cardinoma histology NSCLC. Mixed tumors with be categorized by the predominant cell type. Subjects with mixed small cell lung cancer and NSCLC histology or large cell neuroendocrine carcinoma histology are ineligible. Subjects with sarcomatoid carcinoma are ineligible.
3. The subject is deemed to have unresectable NSCLC by multidisciplinary evaluation that must include a thoracic surgeon who performs lung cancer surgery as a significant part of their practice.
4. Stage IIIB N3 and Stages IIIC, IVA and IVB NSCLC.
5. [*]History or presence of hematological malignancies unless curatively treated with no evidence of disease ≥ 2 years.
6. [*]History of other malignancy with the following exceptions:

   * Treated malignancy with no known active disease present for ≥ 2 years before enrollment and felt to be at low risk for recurrence by the treating physician.
   * Adequately treated non-melanoma skin cancer (basal or squamous cell cancer) or lentigo maligna without evidence of disease.
   * Adequately treated cervical carcinoma in situ without evidence of disease.
   * Adequately treated breast ductal carcinoma in situ without evidence of disease.
   * Prostatic intraepithelial neoplasia without evidence of prostate cancer.
   * Adequately treated urothelial papillary non-invasive carcinoma or carcinoma in situ.
7. Major surgery within 28 days of cycle 1 day 1. In addition, patients with ongoing clinically relevant complications from prior surgery are not eligible and they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
8. [*]Significant cardiovascular disease, such as New York Heart Association cardiac disease (> Class II), myocardial infarction within 6 months prior to cycle 1 day 1, unstable angina or unstable/uncontrolled cardiac arrhythmias. Patients with cardiac arrhythmias that are adequately controlled with medication (for example chronic, rate controlled atrial fibrillation) are potentially eligible if they are deemed to be surgical candidates and do not meet other exclusion criteria. Patients with 1st degree atrioventricular [AV] block or asymptomatic left anterior fascicular block [LAFB/right bundle branch block [RBBB] are eligible.
9. [*]Gastrointestinal (GI ) tract disease causing inability to take oral medication, refractory nausea and vomiting, uncontrolled diarrhea, significant small bowel resection or gastric bypass surgery, use of feeding tubes, malabsorption syndrome, requirement for intravenous alimentation, or uncontrolled inflammatory GI disease (for example Crohn's disease, ulcerative colitis).
10. Infections requiring more than 5 days of parenteral antibiotics, antivirals, or antifungals within 2 weeks prior to cycle 1 day 1. Anti-infective therapy must be completed at least 7 days before cycle 1 day 1. Prophylactic antibiotics are allowed following approval by the trial PI.
11. Previous history of interstitial lung disease or drug-induced pneumonitis.
12. [*]Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
13. [*]Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the treating physician (local principal investigator or sub-investigator)would make the patient inappropriate for entry into the study.
14. Patients with newly diagnosed (as documented by an audiology assessment performed prior to study enrollment) or pre-existing moderate or severe sensorineural hearing loss are not eligible to receive cisplatin but may be treated with carboplatin following discussion of the risks and benefits at the discretion of the treating physician.
15. [*]Current CTCAE version 5.0 grade ≥ 2 peripheral neuropathy.
16. [*]Unwillingness or inability to follow the procedures required in the protocol.
17. [*]Psychological,familial,sociological or geographicalfactors potentially hampering compliance with the study protocol and follow-up schedule.
18. Positive test for hepatitis B virus surface antigen (HBsAg). If the patient is negative for HBsAg) but has positive hepatitis B core antibody, then hepatitis B surface antibody [Anti-HBs] testing is necessary (Hepatitis B core antibody testing is not required for screening but if this is done and is positive, then anti-HBs testing is necessary). Undetectable anti-HBs in this setting would suggest unclear and possible infecition and needs exclusion. Patients receiving antiviral therapy for Hepatitis B or C are not eligible.
19. Positive Hepatitis C virus antibody. In this case hepatitis C virus ribonucleic acid [HCV RNA] is necessary. Detectable HCV RNA indicating acute or chronic infection renders the subject ineligible.
20. [*]Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiencysyndrome.
21. Subject has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmetter-Guerin (BCG) and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg FluMist®) are live attenuated vaccines and are not allowed. Patients who enroll in the clinical protocol should not receive a live vaccine while receiving investigational product and up to 30 days after the last dose of investigational product. 34
22. [*]Regular use of illicit drugs or history (within the past year) of substance abuse (including alcohol).
23. [*]Subject is unwilling to take corticosteroid premedication for pemetrexed.
24. [*]Subject is unwilling or unable to take folic acid or vitamin B12 (intramuscular injection per label) supplementation.
25. [*]Subject is unable or unwilling to interrupt aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs), other than aspirin dose ≤ 1.3gr per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam).
26. Use of known cytochrome P450 (CYP) 3A4 sensitive substrates (with a narrow therapeutic window) or P-gp sensitive substrates (with a narrow therapeutic window) within 14 days or 5 half-lives of the drug or its major active metabolite, whichever is longer, prior to study day 1 that was not reviewed and approved by the principal investigator.
27. Use of strong inducers of CYP3A4 (including herbal supplements such as St. John's wort) within 14 days or 5 half-lives (whichever is longer) prior to study day 1 that was not reviewed and approved by the principal investigator.
28. Use of warfarin. Other anticoagulation may be allowed with PI approval.
29. [*]History of severe hypersensitivity reaction to any component of the study drug treatment (cisplatin/carboplatinpemetrexed, sotorasib).
30. [*]Brain metastatic disease cannot be confidently excluded due to inability to receive both iodinated contrast for CT scans and gadolinium contrast for MRI scans.
31. [*]Female subject who is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment with:

    * Sotorasib and for an additional 7 days after the last dose of sotorasib
    * Cisplatin (or Carboplatin) and Pemetrexed and for an additional 6 months after the last dose of cisplatin/carboplatin or pemetrexed.
32. [*]Female subjects of childbearing potential unwilling to use one highly effective method of contraception (such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner). during treatment with:

    * Sotorasib and for an additional 7 days after the last dose of sotorasib
    * Cisplatin (or Carboplatin) and Pemetrexed and for an additional 6 months after the last dose of cisplatin/carboplatin or pemetrexed.
33. [*]Female subjects of childbearing potential unwilling to use one highly effective method of contraception (such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner). during treatment with:

    * Sotorasib and for an additional 7 days after the last dose of sotorasib.
    * Cisplatin (or Carboplatin) and Pemetrexed and for an additional 6 months after the last dose of cisplatin/carboplatin or pemetrexed. Female subject of childbearing potential is defined as any female who has experienced menarche and who has not undergone surgicalsterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes
34. [*]Female subjects of childbearing potential with a positive pregnancy test assessed at screening or day 1 by a serum pregnancy test and/or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG).
35. [*]Male subjects with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment with:

    * Sotorasib and for an additional 7 days after the last dose of sotorasib.
    * Cisplatin (or Carboplatin) and Pemetrexed and for an additional 3 months after the last dose of cisplatin (or carboplatin) and pemetrexed.
36. [*]Male subjects with a pregnant partner who are unwilling to practice sexual abstinence or use a condom during heterosexual intercourse during treatment with:

    * Sotorasib and for an additional 7 days after the last dose of sotorasib.
    * Cisplatin (or Carboplatin) plus pemetrexed and for an additional 6 months after the last dose of cisplatin (or carboplatin) plus pemetrexed
37. [*]Male subjects unwilling to abstain from donating sperm during treatment and for an additional 6 months after the last dose of cisplatin (or carboplatin) and pemetrexed.
38. Vulnerable populations including prisoners and cognitively impaired adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2027-10-20 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
Patients with surgically resectable KRAS p.G12C-mutant non-squamous NSCLC as assessed by major pathologic response rate in resected tumor specimens | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinandos Skoulidis, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org